CLINICAL TRIAL: NCT04721496
Title: Measuring Velocity and Power on Unstable Push-up: Differences Between Trained and Untrained Population.
Brief Title: Experimental Study Measuring Power and Execution Speed in 44 Athletes in Push-up Exercise.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Moisés Marquina Nieto, Principal Investigator, Universidad Politecnica de Madrid
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Entrenamiento de potencia
Record Dates: First submitted 2020-04-02; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Power
Keywords: Core; Unstable Devices; Suspension Training; Resistance Training; Strength
MeSH Terms: interventions — Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trained (Experimental): Athletes who had at least 2 years of continuous strength training experience, and at least 6 months of training with unstable situations and device
  Interventions: Behavioral: Power and Speed
- Untrained (Experimental): Athletes who had at least 2 years of continuous strength training experience, but no training experience with unstable situations and devices
  Interventions: Behavioral: Power and Speed

INTERVENTIONS:
Behavioral: Power and Speed — Analysis of the power and speed of execution in 6 conditions of increasing instability Situation 1 is stable and basic execution. Condition 6 is the most unstable.
  The participants performed 2 series of 3 repetitions in each of the situations. All the exercises were executed on the same day.

SUMMARY:
Investigation of power and speed in relation to the increasing instability in a group of untrained athletes and a group of expert athletes. In this way, the effectiveness of unstable training for different types of athletes can be tested.

Our hypothesis is that as instability increases there is a gradual decrease in power and speed of execution, but not too relevant in the expert group.

DETAILED DESCRIPTION:
Introduction

Strength training using devices that induce varying degrees of instability is widely practiced in numerous contexts and has been credited with benefits in prevention, rehabilitation and general health. Several studies have found a progressive decrease in power as the degree of instability increases. However, it is not known how mildly unstable situations are affected, nor are the differences between trained and untrained subjects.

The purpose of the present study was to compare the effect of different degrees of instability on power and speed of execution in a push-up or arm-bottoms exercise, in trained and untrained subjects.

Method

Maximum power (MP) and mean power (BP), and maximum speed (MV) and mean propulsive speed (VA) of push-up were analyzed in 44 subjects, 24 untrained (176.38±5.35 cm, 76.38±6.85 kg, 2.5±1.5 months experience) and 20 trained (178.45±5.91 cm, 83.4±21.56 kg, 15.5±5.3 months experience), under six conditions of increasing instability: 1) stable, 2) device in suspension: rings, 3) monopodal, 4) device in suspension: TRX®, 5) with hands-on Bosu® and 6) with hands-on TRX® and feet on Bosu®.

ELIGIBILITY:
Inclusion Criteria:

* 2 years of continuous strength training
* No injuries of any kind within the last year
* Perform a regular push-up exercise
* Having ever used an unstable device

Exclusion Criteria:

* Previous injuries
* Never have used unstable devices
* Newcomers to strength training

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Power | 1 month
  Analysis of the power exercised in the execution of each exercise It was measured with a linear encoder.
Execution Speed | 1 month
  Analysis of the speed exercised in the execution of each exercise It was measured with a linear encoder.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Rivilla, PhD, Study Director — Universidad Politecnica de Madrid; Jorge Lorenzo-Calvo, PhD, Study Director — Universidad Politecnica de Madrid
Locations (1):
- Facultad Ciencias de la Actividad Física y del Deporte, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marquina Nieto M, Rivilla-Garcia J, de la Rubia A, Lorenzo-Calvo J. Assessment of the Speed and Power of Push-Ups Performed on Surfaces with Different Degrees of Instability. Int J Environ Res Public Health. 2022 Oct 22;19(21):13739. doi: 10.3390/ijerph192113739. PMID 36360619